CLINICAL TRIAL: NCT02880891
Title: School and Hospital of Somatology, Peking University
Brief Title: Effects of Splinted or Non-splinted Single-unit Crowns on Marginal Bone-level Alterations Around Implants
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University (Other)
Collaborators: Dentsply Sirona Implants and Consumables (Industry)
Responsible Party: Principal Investigator, Jianzhang Liu, Associate Clinical Professor, Peking University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PKUSSIRB-201520029
Record Dates: First submitted 2016-08-18; First posted 2016-08-26 (Estimated); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Jaw, Edentulous, Partially
MeSH Terms: conditions — Jaw, Edentulous, Partially

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- splinted (Experimental): splinted crown
  Interventions: Procedure: prothetic procedure
- non-splinted (No Intervention): single crown

INTERVENTIONS:
Procedure: prothetic procedure — splinted crown
  Other Names: crown on the implants
  Arms: splinted

SUMMARY:
The microthreaded and platform switched implants could control the stress in the suitable range. The splint would disturb the function. So it is necessary to know whether the splinted single-unit crowns is fit for the adjacent multi-implants.

Outcome variables: Splinted single-unit crowns on one side implants and non-splinted single-unit crowns on the other side Materials and method: 80-100 consecutive implants in at least 20 patients would be included for implant- supported restorations in the posterior maxilla or mandibular. All patients would be in general good health. For every patient, the same posterior teeth had lost on both sides for more than 6 months. All patients were treated by the same qualified surgeon.

Prosthetics procedure would be performed by an experienced prosthodontist. The two sides were allocated to the test or the control group according to the predefined computer-generated randomization table. Clinical evaluations and radiographic analysis were performed by an oral and maxillofacial radiologist who was not aware of the type of Prosthetics technique that was used.

DETAILED DESCRIPTION:
The microthreaded and platform switched implants could control the stress in the suitable range. The splint would disturb the function. So it is necessary to know whether the splinted single-unit crowns is fit for the adjacent multi-implants.

Outcome variables: Splinted single-unit crowns on one side implants and non-splinted single-unit crowns on the other side Materials and method: 80-100 consecutive implants in at least 20 patients would be included for implant- supported restorations in the posterior maxilla or mandibular. All patients would be in general good health. For every patient, the same posterior teeth had lost on both sides for more than 6 months. All patients were treated by the same qualified surgeon.

Prosthetics procedure would be performed by an experienced prosthodontist. The two sides were allocated to the test or the control group according to the predefined computer-generated randomization table. Clinical evaluations and radiographic analysis were performed by an oral and maxillofacial radiologist who was not aware of the type of Prosthetics technique that was used.

ELIGIBILITY:
Inclusion Criteria:

1. All patients would be in general good health.
2. All patients would need for fixed implant-supported prosthesis in the double posterior maxillae or mandibulae (there were at least two corresponding adjacent teeth lost in both sides from the 1st premolar to 2nd molar).
3. The patients could be followed-up for 36 months after prosthetic loading
4. A wide ridge of bone allowing the insertion of a 4mm platform implant and at least 8mm of bone in vertical height would be required.
5. The same posterior teeth had lost on both sides for more than 6 months.

Exclusion Criteria:

1. For implant site, a ridge of bone do not allow the insertion of a 4mm platform implant and at least 8mm of bone in vertical height.
2. Current need for pre-surgical bone or soft tissue augmentation in the planned implant area;
3. Uncontrolled pathologic processes in the oral cavity;
4. History of radiation therapy in the head and neck region;
5. History of chemotherapy within 5 years prior to surgery;
6. Systemic or local disease or condition that could compromise post-operative healing and/or osseointegration;
7. Uncontrolled diabetes mellitus;
8. Corticosteroids or any other medication that could influence post-operative healing and/or osseointegration;
9. Smoking more than 10 cigarettes/day;
10. Present alcohol and/or drug abuse

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-09; Primary Completion 2024-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Marginal Bone Levels (MBL) | three years
  marginal bone level around the implants using CT scan
Probing Pocket Depth (PPD) | three years
  Probing Pocket Depth (PPD) for the implants
Plaque (implant level) | three years
  Plaque (implant level) of the crowns
Bleeding on Probing (Implant level) | three years
  Bleeding on Probing of the crowns

CONTACTS AND LOCATIONS:
Overall Officials: Jianzhang Liu, Doctor, Principal Investigator — Department of Prosthodontics School and Hospital of Stomatology of Peking University
Locations (1):
- Department of Prosthodontics, Peking University School and Hospital of Stomatology, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No